CLINICAL TRIAL: NCT01820455
Title: Methicillin-resistant Staphylococcus Aureus in a Trauma Population: Does Decolonization Prevent Infection?
Brief Title: MRSA in a Trauma Population: Does Decolonization Prevent Infection?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura Brown, Research Coordinator, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTI-TRA-10-020
Record Dates: First submitted 2013-03-20; First posted 2013-03-28 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: MRSA Colonization
Keywords: MRSA decolonization; MRSA subtyping; MRSA infection rates
MeSH Terms: interventions — Chlorhexidine; Mupirocin; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine, Mupirocin (Active Comparator): Chlorhexidine baths and intranasal Mupirocin ointment daily for 5 days
  Interventions: Drug: Chlorhexidine, Mupirocin
- Soap baths, Lubricating jelly (Placebo Comparator): Soap and water baths with lubricating jelly to each nare daily for 5 days
  Interventions: Drug: Soap baths, Lubricating Jelly

INTERVENTIONS:
Drug: Chlorhexidine, Mupirocin — Chlorhexidine baths and intranasal mupirocin ointment once daily for five days
  Other Names: Hibiclens; Bactroban
  Arms: Chlorhexidine, Mupirocin
Drug: Soap baths, Lubricating Jelly — Soap and water baths with lubricating jelly to the nares, once daily for 5 days
  Arms: Soap baths, Lubricating jelly

SUMMARY:
All trauma patients admitted to certain Intensive Care Units (ICU) will have Methicillin-resistant Staphylococcus aureus (MRSA) nasal swabs performed to determine MRSA colonization status. Only those patients who are determined to be colonized with MRSA at admission will be included in the study. All patients must be age 18 and older, admitted directly to the ICU from either the Emergency Department or the operating room with trauma-related injuries, and must not have active or recent known history of MRSA infections. Once patients have been determined to be colonized with MRSA, they will be randomized to receive "decolonization" treatment or placebo. "Decolonization" treatment will include Chlorhexidine baths and Mupirocin ointment to both nares for 5 days and placebo will entail "routine" soap baths and Lubricating Jelly. Both groups will be kept on standard contact precautions throughout the course of the study. Repeat nasal swabs will be performed at the completion of the treatment regimen to determine the efficacy. Patients will be screened for invasive MRSA infections as dictated by their clinical course. The primary outcome measure will be invasive MRSA infection rate (pneumonia, urinary tract infection, bacteremia and soft tissue infection). Secondary endpoints include hospital lengths of stay, ICU lengths of stay, mechanical ventilatory support requirements, colonization status at the end of treatment, and death rates. As determined by our power analysis, we aim to enroll 75 patients in each arm over the course of 12-24 months.

DETAILED DESCRIPTION:
Partway through the enrollment period, it was determined that in the best interests of the patients, the protocol would be altered to eliminate the randomization process and treat all patients with the decolonization treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* colonized with MRSA at admission
* age of 18 years or older
* admitted directly to the ICU from either the ED or the OR with trauma-related injuries

Exclusion Criteria:

* active or recent known history of MRSA infection
* previous institutionalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of patients decolonized following treatment | Up to 24 months
  Measurement of decolonization of MRSA as determined by polymerase chain reaction (PCR) from the nares of critically ill trauma population following treatment.

SECONDARY OUTCOMES:
Number of decolonized patients who develop further infections versus number of infections developed by patients who remain colonized | up to 24 months
  Evaluate the difference between the number of patients who are decolonized following treatment who later develop invasive MRSA infections versus those who remain colonized and develop infections.
Evaluate the genotype and virulence factors of initial colonization and additional MRSA sources | up to 24 months
  Evaluate the genotypes of the initial MRSA sampled and additional sources developed by the patient. This will determine if patients are developing additional infections from outside sources or from the same strain of MRSA with which they were originally colonized.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Maxwell, MD, Principal Investigator — University of Tennessee
Locations (1):
- Erlanger Hospital, Chattanooga, Tennessee, United States

REFERENCES:
- [Background] Croft CA, Mejia VA, Barker DE, Maxwell RA, Dart BW, Smith PW, Burns RP. Methicillin-resistant Staphylococcus aureus in a trauma population: does colonization predict infection? Am Surg. 2009 Jun;75(6):458-61; discussion 461-2. PMID 19545092